CLINICAL TRIAL: NCT04647110
Title: Real-world Study of Non-small Cell Lung Cancer Treatment With ALK-tyrosine Kinase Inhibitors (ALK TKI) in Sweden: Drug Sequencing, Treatment Duration and Overall Survival - A Retrospective Study Using Swedish Register Data
Brief Title: Real-world Therapy of ALK-positive NSCLC in Sweden: the Sequencing of ALK Tyrosine Kinase Inhibitor Drugs and Their Therapeutic Outcomes Based on Data From National Registers.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461035; SEQUIA (Other: Alias Study Number)
Record Dates: First submitted 2020-11-25; First posted 2020-11-30 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: ALK-positive NSCLC
MeSH Terms: interventions — Crizotinib; alectinib; brigatinib; ceritinib; lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Swedish Anaplastic lymphoma kinase (ALK) positive Non-small cell lung cancer (NSCLC) patients
  Interventions: Drug: crizotinib; Drug: alectinib; Drug: brigatinib; Drug: ceritinib; Drug: lorlatinib

INTERVENTIONS:
Drug: crizotinib — as provided in real world practice
Drug: alectinib — as provided in real world practice
Drug: brigatinib — as provided in real world practice
Drug: ceritinib — as provided in real world practice
Drug: lorlatinib — as provided in real world practice

SUMMARY:
This study aims to explore for the first time how the different ALK TKIs have been sequenced in real-world clinical practice and with which outcomes for Swedish lung cancer patients

ELIGIBILITY:
Inclusion Criteria:

-Inclusion criteria for ALK-positive NSCLC patients will be based on prescription data i.e. defines eligible patients as adult patients with at least one filled prescription of ALK-inhibitors identified by the national prescription register. Only prescriptions filled at pharmacies can be captured in prescription registers, as they do not include data on hospital drugs. ALK-inhibitor treatments for patients with NSCLC are given primarily outside of the hospital setting minimizing the selection bias under the inclusion criteria.

Exclusion Criteria:

-not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with ALK TKIs in Sweden between 2012 and 2019, identified via the national prescription register.
Sampling Method: Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Innovations AB, Sollentuna, Sweden

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population included participants aged greater than or equal to 18 years at index date (date of first ALK TKI prescription), with anaplastic lymphoma kinase (ALK)-positive non-small cell lung cancer (NSCLC) who had at least one filled prescription of ALK tyrosine kinase inhibitors (TKI) registered in the Swedish Prescribed Drug Register, between 01-Jan-2012 to 31-Dec-2020. Data of eligible participants were assessed in approximately 3 months of this retrospective observational study.
Pre-assignment Details: According to application sent to ethical counsel for this study, it was pre-planned not to report data for those cohorts/groups which had less than (<) 5 participants at the index date. Hence, due to ethical compliance study team ensured results would only be displayed on an aggregate level for reporting arms having greater than or equal to (>=) 5 participants at index date.
Groups:
- Participants With No First Line Chemotherapy: Participants included in this arm received at least one filled prescription of ALK TKIs in real world practices, with no first line chemotherapy treatment. ALK TKIs were crizotinib, alectinib, brigatinib, ceritinib, or lorlatinib.
- Participants With First Line Chemotherapy: Participants included in this arm received at least one filled prescription of ALK TKIs in real world practices, along with first line chemotherapy treatment. ALK TKIs were crizotinib, alectinib, brigatinib, ceritinib, or lorlatinib.
Period: Overall Study
Arm/Group | Participants With No First Line Chemotherapy | Participants With First Line Chemotherapy
Started | 345 | 204
Completed | 345 | 204
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With No First Line Chemotherapy | Participants With First Line Chemotherapy | Total
Number analyzed (Participants) | 345 | 204 | 549
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.08 (13.96) | 63.24 (13.28) | 63.13 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 112 | 301
  Male | 156 | 92 | 248
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Secondary Outcome: Duration of Treatment: Based on Treatment Cohort Groups
Description: Duration of treatment was defined as number of days on treatment calculated based on pharmaceutical specialties in Sweden (FASS) recommended dose for filled prescriptions of ALK-inhibitors taking permissible gap and stockpiling into account. Results were reported for treatment cohort groups based on generation of ALK treatment and were as following: Group A1 = chemotherapy + crizotinib (first generation ALK TKI) + any second (2nd) generation ALK TKI; Group A2 = crizotinib + any 2nd generation ALK TKI; Group B1: chemotherapy + crizotinib + any 2nd generation ALK TKI + any other 2nd generation ALK TKI; Group B2 = crizotinib + any 2nd generation ALK TKI + any other 2nd generation ALK TKI; Group C1 = chemotherapy + crizotinib + any 2nd generation ALK TKI + lorlatinib (third generation ALK TKI); Group C2: crizotinib + any 2nd generation ALK TKI + lorlatinib and Group D1 = any 2nd generation ALK TKI + any other 2nd generation ALK TKI.
Time Frame: From index date to treatment completion/discontinuation during data identification period of 9 years (retrieved data assessed in this observational study for approximately 3 months)
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure based on generation of ALK treatment.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Group A1: Participants included in this arm received chemotherapy, crizotinib, and any second generation ALK TKI, in real world practices. Second generation ALK TKIs considered were alectinib, brigatinib, or ceritinib.
- Group A2: Participants included in this arm received crizotinib and any second generation ALK TKI in real world practices. Second generation ALK TKIs considered were alectinib, brigatinib, or ceritinib.
- Group B1: Participants included in this arm received chemotherapy, crizotinib and any two second generation ALK TKIs in real world practices. Second generation ALK TKIs considered were alectinib, brigatinib, or ceritinib.
- Group B2: Participants included in this arm received, crizotinib and any two second generation ALK TKIs in real world practices. Second generation ALK TKIs considered were alectinib, brigatinib, or ceritinib.
- Group C1: Participants included in this arm received chemotherapy, crizotinib, any second generation ALK TKI and lorlatinib in real world practices. Second generation ALK TKIs considered were alectinib, brigatinib, or ceritinib.
- Group C2: Participants included in this arm received crizotinib, any second generation ALK TKI and lorlatinib in real world practices. Second generation ALK TKIs considered were alectinib, brigatinib, or ceritinib.
- Group D1: Participants included in this arm received any two second generation ALK TKIs in real world practices. Second generation ALK TKIs considered were alectinib, brigatinib, or ceritinib.
Arm/Group | Group A1 | Group A2 | Group B1 | Group B2 | Group C1 | Group C2 | Group D1
Number analyzed (Participants) | 29 | 71 | 10 | 14 | 5 | 9 | 9
Years | 1.66 (1.28) | 1.86 (1.31) | 3.37 (1.24) | 2.45 (1.53) | 2.56 (1.42) | 2.72 (1.03) | 1.36 (0.75)

2. Secondary Outcome: Duration of Treatment: Based on Chemotherapy Status
Description: Duration of treatment was defined as number of days on treatment calculated based on pharmaceutical specialties in Sweden (FASS) recommended dose for filled prescriptions of ALK-inhibitors taking permissible gap and stockpiling into account. Results were reported based on chemotherapy status.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Participants With No First Line Chemotherapy | Participants With First Line Chemotherapy
Number analyzed (Participants) | 345 | 204
Years | 1.23 (1.28) | 1.07 (1.28)

3. Secondary Outcome: Duration of Treatment: Based on ALK Sequencing, 1 Line of ALK TKI Treatment
Description: Duration of treatment was defined as number of days on treatment calculated based on FASS recommended dose for filled prescriptions of ALK-inhibitors taking permissible gap and stockpiling into account. Reporting arms were based on type of ALK TKI, with or without chemotherapy. ALK TKIs considered were crizotinib, alectinib, ceritinib.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed (N)" signifies participants evaluable for this measure and received only 1 line of ALK TKIs with/ without chemotherapy. Due to ethical compliance, it was pre-planned not to report data for those reporting groups which had <5 participants at the index date.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Crizotinib: Participants included in this arm received only crizotinib in real world practices
- Alectinib: Participants included in this arm received only alectinib in real world practices.
- Ceritinib: Participants included in this arm received only ceritinib in real world practices.
- Crizotinib + Chemotherapy: Participants included in this arm received crizotinib in real world practices along with chemotherapy.
- Alectinib + Chemotherapy: Participants included in this arm received alectinib in real world practices along with chemotherapy.
- Ceritinib + Chemotherapy: Participants included in this arm received ceritinib in real world practices along with chemotherapy.
Arm/Group | Crizotinib | Alectinib | Ceritinib | Crizotinib + Chemotherapy | Alectinib + Chemotherapy | Ceritinib + Chemotherapy
Number analyzed (Participants) | 116 | 105 | 4 | 95 | 41 | 5
Years
  First Line ALK TKI Treatment Duration | 0.72 (1.19) | 0.92 (0.82) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.50 (0.80) | 0.80 (0.88) | 1.01 (1.23)
  Total Sequence Treatment Duration | 0.72 (1.19) | 0.92 (0.82) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.50 (0.80) | 0.80 (0.88) | 1.01 (1.23)

4. Secondary Outcome: Duration of Treatment: Based on ALK Sequencing, 2 Lines of ALK TKI Treatment
Description: Duration of treatment was defined as number of days on treatment calculated based on FASS recommended dose for filled prescriptions of ALK-inhibitors taking permissible gap and stockpiling into account. Reporting arms were based on type of first line ALK TKI treatment, and second line of ALK TKI treatment, with or without chemotherapy.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. "Overall Number of Participants Analyzed (N)": participants evaluable for this measure and received only 2 lines of ALK TKIs with/ without chemotherapy. Groups with "N" =0: no participants with respective ALK TKI sequencing. Due to ethical compliance, it was pre-planned not to report data for those reporting groups which had <5 participants at the index date.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Crizotinib + Alectinib: Participants included in this arm received crizotinib as first line ALK KI treatment and alectinib as second line ALK TKI treatment, in real world practices.
- Crizotinib + Brigatinib: Participants included in this arm received crizotinib as first line ALK KI treatment and brigatinib as second line ALK TKI treatment, in real world practices.
- Crizotinib + Ceritinib: Participants included in this arm received crizotinib as first line ALK KI treatment and ceritinib as second line ALK TKI treatment, in real world practices.
- Alectinib + Brigatinib: Participants included in this arm received alectinib as first line ALK KI treatment and brigatinib as second line ALK TKI treatment, in real world practices.
- Alectinib + Ceritinib: Participants included in this arm received alectinib as first line ALK KI treatment and ceritinib as second line ALK TKI treatment, in real world practices.
- Alectinib + Lorlatinib: Participants included in this arm received alectinib as first line ALK KI treatment and lorlatinib as second line ALK TKI treatment, in real world practices.
- Ceritinib + Alectinib: Participants included in this arm received ceritinib as first line ALK KI treatment and alectinib as second line ALK TKI treatment, in real world practices.
- Ceritinib + Brigatinib: Participants included in this arm received ceritinib as first line ALK KI treatment and brigatinib as second line ALK TKI treatment, in real world practices.
- Ceritinib + Lorlatinib: Participants included in this arm received ceritinib as first line ALK KI treatment and lorlatinib as second line ALK TKI treatment, in real world practices.
- Crizotinib + Alectinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK KI treatment and alectinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Brigatinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK KI treatment and brigatinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Ceritinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK KI treatment and ceritinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Alectinib + Brigatinib + Chemotherapy: Participants included in this arm received alectinib as first line ALK KI treatment and brigatinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Alectinib + Ceritinib + Chemotherapy: Participants included in this arm received alectinib as first line ALK KI treatment and ceritinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Alectinib + Lorlatinib + Chemotherapy: Participants included in this arm received alectinib as first line ALK KI treatment and lorlatinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Ceritinib + Alectinib + Chemotherapy: Participants included in this arm received ceritinib as first line ALK KI treatment and alectinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Ceritinib + Brigatinib + Chemotherapy: Participants included in this arm received ceritinib as first line ALK KI treatment and brigatinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
- Ceritinib + Lorlatinib + Chemotherapy: Participants included in this arm received ceritinib as first line ALK KI treatment and lorlatinib as second line ALK TKI treatment, in real world practices along with chemotherapy.
Arm/Group | Crizotinib + Alectinib | Crizotinib + Brigatinib | Crizotinib + Ceritinib | Alectinib + Brigatinib | Alectinib + Ceritinib | Alectinib + Lorlatinib | Ceritinib + Alectinib | Ceritinib + Brigatinib | Ceritinib + Lorlatinib | Crizotinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Chemotherapy | Alectinib + Brigatinib + Chemotherapy | Alectinib + Ceritinib + Chemotherapy | Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Chemotherapy | Ceritinib + Brigatinib + Chemotherapy | Ceritinib + Lorlatinib + Chemotherapy
Number analyzed (Participants) | 33 | 0 | 38 | 8 | 0 | 6 | 1 | 0 | 1 | 9 | 2 | 18 | 2 | 1 | 7 | 2 | 0 | 0
Years
  First Line ALK TKI Treatment Duration | 1.01 (0.80) |  | 0.62 (0.45) | 0.61 (0.51) |  | 0.95 (0.62) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 1.42 (1.31) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.81 (0.70) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.50 (0.60) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |
  Second Line ALK TKI Treatment Duration | 1.62 (1.07) |  | 0.58 (0.72) | 0.55 (0.34) |  | 0.27 (0.23) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.75 (0.89) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.37 (0.67) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.40 (0.37) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |
  Total Sequence Treatment Duration | 2.62 (1.33) |  | 1.21 (0.86) | 1.16 (0.51) |  | 1.22 (0.57) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 2.17 (1.32) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 1.18 (0.99) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.89 (0.64) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |

5. Secondary Outcome: Duration of Treatment: Based on ALK Sequencing, 3 Lines of ALK TKI Treatment
Description: Duration of treatment was defined as number of days on treatment calculated based on FASS recommended dose for filled prescriptions of ALK-inhibitors taking permissible gap and stockpiling into account. Reporting arms were based on type of first line ALK TKI treatment, second line of ALK TKI treatment, and third line of ALK TKI treatment with or without chemotherapy.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. "Overall Number of Participants Analyzed (N)": participants evaluable for this measure and received only 3 lines of ALK TKIs with/ without chemotherapy. Groups with "N" =0: no participants with respective ALK TKI sequencing. Due to ethical compliance, it was pre-planned not to report data for those reporting groups which had <5 participants at the index date.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Crizotinib + Alectinib + Ceritinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment and ceritinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Alectinib + Lorlatinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment and lorlatinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Alectinib + Brigatinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment and brigatinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Ceritinib + Alectinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, ceritinib as second line ALK TKI treatment and alectinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Ceritinib + Lorlatinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, ceritinib as second line ALK TKI treatment and lorlatinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Ceritinib + Brigatinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, ceritinib as second line ALK TKI treatment and brigatinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Brigatinib + Alectinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, brigatinib as second line ALK TKI treatment and alectinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Brigatinib + Lorlatinib: Participants included in this arm received crizotinib as first line ALK TKI treatment, brigatinib as second line ALK TKI treatment and lorlatinib as third line ALK TKI treatment, in real world practices.
- Alectinib + Brigatinib + Lorlatinib: Participants included in this arm received alectinib as first line ALK TKI treatment, brigatinib as second line ALK TKI treatment and lorlatinib as third line ALK TKI treatment, in real world practices.
- Alectinib + Lorlatinib + Brigatinib: Participants included in this arm received alectinib as first line ALK TKI treatment, lorlatinib as second line ALK TKI treatment and brigatinib as third line ALK TKI treatment, in real world practices.
- Alectinib + Lorlatinib + Ceritinib: Participants included in this arm received alectinib as first line ALK TKI treatment, lorlatinib as second line ALK TKI treatment and ceritinib as third line ALK TKI treatment, in real world practices.
- Ceritinib + Alectinib + Lorlatinib: Participants included in this arm received ceritinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment and lorlatinib as third line ALK TKI treatment, in real world practices.
- Ceritinib + Alectinib + Brigatinib: Participants included in this arm received ceritinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment and brigatinib as third line ALK TKI treatment, in real world practices.
- Crizotinib + Alectinib + Ceritinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment, ceritinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Alectinib + Lorlatinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment, lorlatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Alectinib + Brigatinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment, brigatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Ceritinib + Alectinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, ceritinib as second line ALK TKI treatment, alectinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Ceritinib + Lorlatinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, ceritinib as second line ALK TKI treatment, lorlatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Ceritinib + Brigatinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, ceritinib as second line ALK TKI treatment, brigatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Brigatinib + Alectinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, brigatinib as second line ALK TKI treatment, alectinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Crizotinib + Brigatinib + Lorlatinib + Chemotherapy: Participants included in this arm received crizotinib as first line ALK TKI treatment, brigatinib as second line ALK TKI treatment, lorlatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Alectinib + Brigatinib + Lorlatinib + Chemotherapy: Participants included in this arm received alectinib as first line ALK TKI treatment, brigatinib as second line ALK TKI treatment, lorlatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Alectinib + Lorlatinib + Brigatinib + Chemotherapy: Participants included in this arm received alectinib as first line ALK TKI treatment, lorlatinib as second line ALK TKI treatment, brigatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Alectinib + Lorlatinib + Ceritinib + Chemotherapy: Participants included in this arm received alectinib as first line ALK TKI treatment, lorlatinib as second line ALK TKI treatment, ceritinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Ceritinib + Alectinib + Lorlatinib + Chemotherapy: Participants included in this arm received ceritinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment, lorlatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
- Ceritinib + Alectinib + Brigatinib + Chemotherapy: Participants included in this arm received ceritinib as first line ALK TKI treatment, alectinib as second line ALK TKI treatment, brigatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
Arm/Group | Crizotinib + Alectinib + Ceritinib | Crizotinib + Alectinib + Lorlatinib | Crizotinib + Alectinib + Brigatinib | Crizotinib + Ceritinib + Alectinib | Crizotinib + Ceritinib + Lorlatinib | Crizotinib + Ceritinib + Brigatinib | Crizotinib + Brigatinib + Alectinib | Crizotinib + Brigatinib + Lorlatinib | Alectinib + Brigatinib + Lorlatinib | Alectinib + Lorlatinib + Brigatinib | Alectinib + Lorlatinib + Ceritinib | Ceritinib + Alectinib + Lorlatinib | Ceritinib + Alectinib + Brigatinib | Crizotinib + Alectinib + Ceritinib + Chemotherapy | Crizotinib + Alectinib + Lorlatinib + Chemotherapy | Crizotinib + Alectinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Alectinib + Chemotherapy | Crizotinib + Ceritinib + Lorlatinib + Chemotherapy | Crizotinib + Ceritinib + Brigatinib + Chemotherapy | Crizotinib + Brigatinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Lorlatinib + Chemotherapy | Alectinib + Brigatinib + Lorlatinib + Chemotherapy | Alectinib + Lorlatinib + Brigatinib + Chemotherapy | Alectinib + Lorlatinib + Ceritinib + Chemotherapy | Ceritinib + Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Brigatinib + Chemotherapy
Number analyzed (Participants) | 0 | 7 | 3 | 11 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 6 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Years
  First Line ALK TKI Treatment Duration |  | 1.12 (1.13) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.70 (0.38) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 1.12 (0.63) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  |  |
  Second Line ALK TKI Treatment Duration |  | 1.29 (0.69) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.85 (0.81) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 1.53 (1.31) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  |  |
  Third Line ALK TKI Treatment Duration |  | 0.47 (0.37) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.85 (0.90) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.68 (1.07) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  |  |
  Total Sequence Treatment Duration |  | 2.88 (1.13) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 2.39 (1.65) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 3.34 (1.01) | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA (NA) — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  |  |

6. Secondary Outcome: Duration of Treatment: Based on ALK Sequencing, More Than or Equal to (>=) 4 Lines of ALK TKI Treatment
Description: Duration of treatment was defined as number of days on treatment calculated based on FASS recommended dose for filled prescriptions of ALK-inhibitors taking permissible gap and stockpiling into account. In this outcome measure, duration of treatment was reported for participants who received >=4 lines of ALK inhibitor treatment, with or without chemotherapy.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and received >= 4 lines of ALK TKI treatment with or without chemotherapy.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- >=4 Lines of ALK TKI: Participants included in this arm received at least 4 different ALK TKIs, in real world practices.
- >=4 Lines of ALK TKI With Chemotherapy: Participants included in this arm received at least 4 different ALK TKIs, in real world practices along with chemotherapy.
Arm/Group | >=4 Lines of ALK TKI | >=4 Lines of ALK TKI With Chemotherapy
Number analyzed (Participants) | 8 | 7
Years
  First Line ALK TKI Treatment Duration | 1.09 (0.61) | 1.56 (0.82)
  Second Line ALK TKI Treatment Duration | 1.01 (0.73) | 0.73 (0.49)
  Third Line ALK TKI Treatment Duration | 0.80 (0.63) | 0.63 (0.56)
  Fourth Line ALK TKI Treatment Duration | 0.52 (0.48) | 0.47 (0.50)
  Total Sequence Treatment Duration | 3.42 (0.98) | 3.40 (1.76)

7. Primary Outcome: Overall Survival (OS): Based on Treatment Cohort Groups
Description: OS was defined as the time from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data). Kaplan-Meier method was used for analysis. Results were reported for treatment cohort groups based on generation of ALK treatment and were as following: Group A1 = chemotherapy + crizotinib (first generation ALK TKI) + any second (2nd) generation ALK TKI; Group A2 = crizotinib + any 2nd generation ALK TKI; Group B1: chemotherapy + crizotinib + any 2nd generation ALK TKI + any other 2nd generation ALK TKI; Group B2 = crizotinib + any 2nd generation ALK TKI + any other 2nd generation ALK TKI; Group C1 = chemotherapy + crizotinib + any 2nd generation ALK TKI + lorlatinib (third generation ALK TKI); Group C2: crizotinib + any 2nd generation ALK TKI + lorlatinib and Group D1 = any 2nd generation ALK TKI + any other 2nd generation ALK TKI.
Time Frame: From index date to the date of death due to any cause or censoring date, during data identification period of 9 years (retrieved data assessed in this observational study for approximately 3 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Group A1 | Group A2 | Group B1 | Group B2 | Group C1 | Group C2 | Group D1
Number analyzed (Participants) | 29 | 71 | 10 | 14 | 5 | 9 | 9
Years | 1.94 [1.22 to 3.35] | 2.30 [1.67 to 3.02] | 4.56 [2.41 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event. | 2.94 [2.07 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. | 5.41 [NA to NA] — Upper and lower limit for 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event.

8. Primary Outcome: Overall Survival: Based on Chemotherapy Status
Description: OS was defined as the time from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data). Kaplan-Meier method was used for analysis. Results were reported based on chemotherapy status.
Time Frame: as for outcome 7
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Participants With No First Line Chemotherapy | Participants With First Line Chemotherapy
Number analyzed (Participants) | 345 | 204
Years | 2.02 [1.60 to 2.58] | 1.44 [0.89 to 1.98]

9. Primary Outcome: Overall Survival: Based on Central Nervous System (CNS) Metastases Status
Description: OS was defined as the time from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data). Kaplan-Meier method was used for analysis. In this outcome measure, participants were grouped on basis of their CNS-metastases status.
Time Frame: as for outcome 7
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Years
Groups:
- Participants With No CNS Metastases: Participants included in this arm received at least one filled prescription of ALK TKIs in real world practices, with or without first line chemotherapy treatment and had no CNS metastases during 2 years period prior to index date. ALK TKIs were crizotinib, alectinib, brigatinib, ceritinib, or lorlatinib
- Participants With CNS Metastases: Participants included in this arm received at least one filled prescription of ALK TKIs in real world practices, with or without first line chemotherapy treatment and had CNS metastases during 2 years period prior to index date. ALK TKIs were crizotinib, alectinib, brigatinib, ceritinib, or lorlatinib.
Arm/Group | Participants With No CNS Metastases | Participants With CNS Metastases
Number analyzed (Participants) | 520 | 29
Years | 1.94 [1.52 to 2.26] | 0.61 [0.34 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event.

10. Primary Outcome: Overall Survival: Based on ALK Sequencing, 1 Line of ALK TKI Treatment
Description: OS was defined as the time from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data). Kaplan-Meier method was used for analysis. In this outcome measure, OS was reported for participants who received 1 line of ALK TKI treatment. Reporting arms were based on type of ALK TKI, with or without chemotherapy. ALK TKIs considered were crizotinib, alectinib, ceritinib.
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Crizotinib | Alectinib | Ceritinib | Crizotinib + Chemotherapy | Alectinib + Chemotherapy | Ceritinib + Chemotherapy
Number analyzed (Participants) | 116 | 105 | 4 | 95 | 41 | 5
Years | 0.88 [0.60 to 1.08] | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 0.63 [0.46 to 0.78] | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. | 0.59 [0.44 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event.

11. Primary Outcome: Overall Survival: Based on ALK Sequencing, 2 Lines of ALK TKI Treatment
Description: OS was defined as the time from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data). Kaplan-Meier method was used for analysis. In this outcome measure OS was reported for participants who received 2 lines of ALK TKI treatment. Reporting arms were based on type of first line ALK TKI treatment and second line of ALK TKI treatment, with or without chemotherapy.
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Crizotinib + Alectinib | Crizotinib + Brigatinib | Crizotinib + Ceritinib | Alectinib + Brigatinib | Alectinib + Ceritinib | Alectinib + Lorlatinib | Ceritinib + Alectinib | Ceritinib + Brigatinib | Ceritinib + Lorlatinib | Crizotinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Chemotherapy | Alectinib + Brigatinib + Chemotherapy | Alectinib + Ceritinib + Chemotherapy | Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Chemotherapy | Ceritinib + Brigatinib + Chemotherapy | Ceritinib + Lorlatinib + Chemotherapy
Number analyzed (Participants) | 33 | 0 | 38 | 8 | 0 | 6 | 1 | 0 | 1 | 9 | 2 | 18 | 2 | 1 | 7 | 2 | 0 | 0
Years | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. |  | 1.27 [1.14 to 1.94] | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. |  | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 2.69 [1.22 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 1.38 [0.76 to 2.94] | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |

12. Primary Outcome: Overall Survival: Based on ALK Sequencing, 3 Lines of ALK TKI Treatment
Description: OS was defined as the time from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data). Kaplan-Meier method was used for analysis. In this outcome measure OS was reported for participants who received 3 lines of ALK inhibitor treatment. Reporting arms were based on type of first line ALK TKI treatment, second line of ALK TKI treatment and third line of ALK TKI treatment with or without, chemotherapy.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Years
Groups:
- Alectinib + Lorlatinib + Brigatinib +Chemotherapy: Participants included in this arm received alectinib as first line ALK TKI treatment, lorlatinib as second line ALK TKI treatment, brigatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
Arm/Group | Crizotinib + Alectinib + Ceritinib | Crizotinib + Alectinib + Lorlatinib | Crizotinib + Alectinib + Brigatinib | Crizotinib + Ceritinib + Alectinib | Crizotinib + Ceritinib + Lorlatinib | Crizotinib + Ceritinib + Brigatinib | Crizotinib + Brigatinib + Alectinib | Crizotinib + Brigatinib + Lorlatinib | Alectinib + Brigatinib + Lorlatinib | Alectinib + Lorlatinib + Brigatinib | Alectinib + Lorlatinib + Ceritinib | Ceritinib + Alectinib + Lorlatinib | Ceritinib + Alectinib + Brigatinib | Crizotinib + Alectinib + Ceritinib + Chemotherapy | Crizotinib + Alectinib + Lorlatinib + Chemotherapy | Crizotinib + Alectinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Alectinib + Chemotherapy | Crizotinib + Ceritinib + Lorlatinib + Chemotherapy | Crizotinib + Ceritinib + Brigatinib + Chemotherapy | Crizotinib + Brigatinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Lorlatinib + Chemotherapy | Alectinib + Brigatinib + Lorlatinib + Chemotherapy | Alectinib + Lorlatinib + Brigatinib +Chemotherapy | Alectinib + Lorlatinib + Ceritinib + Chemotherapy | Ceritinib + Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Brigatinib + Chemotherapy
Number analyzed (Participants) | 0 | 7 | 3 | 11 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 6 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Years |  | 5.41 [NA to NA] — Upper and lower limit for 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 2.78 [2.07 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. | 4.06 [2.41 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  | NA [NA to NA] — Due to ethical compliance data is not reported for reporting arms with <5 participants at index date. |  |  |  |  |

13. Primary Outcome: Overall Survival: Based on ALK Sequencing, More Than or Equal to (>=) 4 Lines of ALK TKI Treatment
Description: OS was defined as the time from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data). Kaplan-Meier method was used for analysis. In this outcome measure, OS was reported for participants who received >=4 lines of ALK inhibitor treatment with or without chemotherapy.
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | >=4 Lines of ALK TKI | >=4 Lines of ALK TKI With Chemotherapy
Number analyzed (Participants) | 8 | 7
Years | 5.49 [3.79 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants. | 5.27 [3.02 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants.

14. Primary Outcome: Percentage of Participants Alive After 5 Years From Index Date: Based on Treatment Cohort Groups
Description: Results were reported for treatment cohort groups based on generation of ALK treatment and were as following: Group A1 = chemotherapy + crizotinib (first generation ALK TKI) + any second (2nd) generation ALK TKI; Group A2 = crizotinib + any 2nd generation ALK TKI; Group B1: chemotherapy + crizotinib + any 2nd generation ALK TKI + any other 2nd generation ALK TKI; Group B2 = crizotinib + any 2nd generation ALK TKI + any other 2nd generation ALK TKI; Group C1 = chemotherapy + crizotinib + any 2nd generation ALK TKI + lorlatinib (third generation ALK TKI); Group C2: crizotinib + any 2nd generation ALK TKI + lorlatinib and Group D1 = any 2nd generation ALK TKI + any other 2nd generation ALK TKI.
Time Frame: 5 years post index date during data identification period of 9 years (retrieved data assessed in this observational study for approximately 3 months)
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed (N)" signifies participants who evaluable for this measure with a follow up of 5 years post index date. Reporting groups with "N" =0 signifies that no participant had a follow up of 5 years post index date.
Measure: Number; unit: Percentage of participants
Arm/Group | Group A1 | Group A2 | Group B1 | Group B2 | Group C1 | Group C2 | Group D1
Number analyzed (Participants) | 16 | 21 | 5 | 2 | 3 | 1 | 0
Percentage of participants | 6.25 | 9.52 | 40.00 | 50.00 | 66.67 | 100 |

15. Primary Outcome: Percentage of Participants Alive After 5 Years From Index Date: Based on Chemotherapy Status
Description: Participants alive after five years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported in this outcome measure. Results were reported based on chemotherapy status.
Time Frame: as for outcome 14
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure with a follow up of 5 years post index date.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With No First Line Chemotherapy | Participants With First Line Chemotherapy
Number analyzed (Participants) | 61 | 61
Percentage of participants | 16.39 | 16.39

16. Primary Outcome: Percentage of Participants Alive After 5 Years From Index Date: Based on CNS Metastases Status
Description: Participants alive after five years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported in this outcome measure. Results were reported based on CNS metastases status.
Time Frame: as for outcome 14
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With No CNS Metastases | Participants With CNS Metastases
Number analyzed (Participants) | 116 | 6
Percentage of participants | 17.24 | 0.00

17. Primary Outcome: Percentage of Participants Alive After 5 Years From Index Date: Based on ALK Sequencing, 1 Line of ALK TKI Treatment
Description: Participants alive after five years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure, participants who received 1 line of ALK TKI treatment, were reported. Reporting arms were based on type of first line ALK TKI treatment, with or without chemotherapy. ALK TKIs considered were crizotinib, alectinib, ceritinib.
Time Frame: as for outcome 14
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure with a follow up of 5 years post index date. Reporting arm with "Overall Number of Participants Analyzed" = 0, signifies that no participant had a follow up of 5 years post index date.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib | Alectinib | Ceritinib | Crizotinib + Chemotherapy | Alectinib + Chemotherapy | Ceritinib + Chemotherapy
Number analyzed (Participants) | 35 | 0 | 0 | 32 | 0 | 0
Percentage of participants | 11.43 |  |  | 0.00 |  |

18. Primary Outcome: Percentage of Participants Alive After 5 Years From Index Date: Based on ALK Sequencing, 2 Lines of ALK TKI Treatment
Description: Participants alive after five years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure, participants who received 2 lines of ALK TKI treatment, were reported. Reporting arms were based on type of first line ALK TKI treatment and second line of ALK TKI treatment, with or without chemotherapy.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib + Alectinib | Crizotinib + Brigatinib | Crizotinib + Ceritinib | Alectinib + Brigatinib | Alectinib + Ceritinib | Alectinib + Lorlatinib | Ceritinib + Alectinib | Ceritinib + Brigatinib | Ceritinib + Lorlatinib | Crizotinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Chemotherapy | Alectinib + Brigatinib + Chemotherapy | Alectinib + Ceritinib + Chemotherapy | Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Chemotherapy | Ceritinib + Brigatinib + Chemotherapy | Ceritinib + Lorlatinib + Chemotherapy
Number analyzed (Participants) | 3 | 0 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of participants | 66.67 |  | 0.00 |  |  |  |  |  |  | 0.00 |  | 7.14 |  |  |  |  |  |

19. Primary Outcome: Percentage of Participants Alive After 5 Years From Index Date: Based on ALK Sequencing, 3 Lines of ALK TKI Treatment
Description: Participants alive after five years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure, participants who received 3 lines of ALK TKI treatment. Reporting arms were based on type of first line ALK TKI treatment, second line of ALK TKI treatment, and third line of ALK TKI treatment, with or without chemotherapy.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Groups:
- Alectinib + Brigatinib + Lorlatinib +Chemotherapy: Participants included in this arm received alectinib as first line ALK TKI treatment, brigatinib as second line ALK TKI treatment, lorlatinib as third line ALK TKI treatment, in real world practices along with chemotherapy.
Arm/Group | Crizotinib + Alectinib + Ceritinib | Crizotinib + Alectinib + Lorlatinib | Crizotinib + Alectinib + Brigatinib | Crizotinib + Ceritinib + Alectinib | Crizotinib + Ceritinib + Lorlatinib | Crizotinib + Ceritinib + Brigatinib | Crizotinib + Brigatinib + Alectinib | Crizotinib + Brigatinib + Lorlatinib | Alectinib + Brigatinib + Lorlatinib | Alectinib + Lorlatinib + Brigatinib | Alectinib + Lorlatinib + Ceritinib | Ceritinib + Alectinib + Lorlatinib | Ceritinib + Alectinib + Brigatinib | Crizotinib + Alectinib + Ceritinib + Chemotherapy | Crizotinib + Alectinib + Lorlatinib + Chemotherapy | Crizotinib + Alectinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Alectinib + Chemotherapy | Crizotinib + Ceritinib + Lorlatinib + Chemotherapy | Crizotinib + Ceritinib + Brigatinib + Chemotherapy | Crizotinib + Brigatinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Lorlatinib + Chemotherapy | Alectinib + Brigatinib + Lorlatinib +Chemotherapy | Alectinib + Lorlatinib + Brigatinib +Chemotherapy | Alectinib + Lorlatinib + Ceritinib + Chemotherapy | Ceritinib + Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Brigatinib + Chemotherapy
Number analyzed (Participants) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of participants |  | 100.00 |  | 50.00 |  |  |  |  |  |  |  |  |  |  |  |  | 25.00 |  |  |  |  |  |  |  |  |

20. Primary Outcome: Percentage of Participants Alive After 5 Years From Index Date: Based on ALK Sequencing, More Than or Equal to (>=) 4 Lines of ALK TKI Treatment
Description: Participants alive after five years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure, data is reported for participants who received >=4 lines of ALK inhibitor treatment with or without chemotherapy.
Time Frame: as for outcome 14
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | >=4 Lines of ALK TKI | >=4 Lines of ALK TKI With Chemotherapy
Number analyzed (Participants) | 2 | 5
Percentage of participants | 100.00 | 100.00

21. Primary Outcome: Percentage of Participants Alive After 6 Years From Index Date: Based on Treatment Cohort Groups
Description: as for outcome 14
Time Frame: 6 years post index date during data identification period of 9 years (retrieved data assessed in this observational study for approximately 3 months)
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed (N)" signifies participants who evaluable for this measure with a follow up of 6 years post index date. Reporting groups with "N" =0 signifies that no participant had a follow up of 6 years post index date.
Measure: Number; unit: Percentage of participants
Arm/Group | Group A1 | Group A2 | Group B1 | Group B2 | Group C1 | Group C2 | Group D1
Number analyzed (Participants) | 5 | 3 | 1 | 0 | 1 | 0 | 0
Percentage of participants | 0.00 | 0.00 | 0.00 |  | 0.00 |  |

22. Primary Outcome: Percentage of Participants Alive After 6 Years From Index Date: Based on Chemotherapy Status
Description: Participants alive after six years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported in this outcome measure. Results were reported based on chemotherapy status.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure with a follow up of 6 years post index date.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With No First Line Chemotherapy | Participants With First Line Chemotherapy
Number analyzed (Participants) | 20 | 26
Percentage of participants | 10.00 | 3.85

23. Primary Outcome: Percentage of Participants Alive After 6 Years From Index Date: Based on CNS Metastases Status
Description: Participants alive after six years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported in this outcome measure. Results were reported based on CNS metastases status.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With No CNS Metastases | Participants With CNS Metastases
Number analyzed (Participants) | 44 | 2
Percentage of participants | 6.82 | 0.00

24. Primary Outcome: Percentage of Participants Alive After 6 Years From Index Date: Based on ALK Sequencing, 1 Line of ALK TKI Treatment
Description: Participants alive after six years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure, participants who received 1 line of ALK TKI treatment, were reported. Reporting arms were based on type of first line ALK TKI treatment, with or without chemotherapy. ALK TKIs considered were crizotinib, alectinib, ceritinib.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data were retrieved from Swedish administrative registers and assessed. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure with a follow up of 6 years post index date. Reporting arm with "Overall Number of Participants Analyzed" = 0, signifies that no participant had a follow up of 6 years post index date.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib | Alectinib | Ceritinib | Crizotinib + Chemotherapy | Alectinib + Chemotherapy | Ceritinib + Chemotherapy
Number analyzed (Participants) | 16 | 0 | 0 | 16 | 0 | 0
Percentage of participants | 12.50 |  |  | 0.00 |  |

25. Primary Outcome: Percentage of Participants Alive After 6 Years From Index Date: Based on ALK Sequencing, 2 Lines of ALK TKI Treatment
Description: Participants alive after six years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure, participants who received 2 lines of ALK TKI treatment, were reported. Reporting arms were based on type of first line ALK TKI treatment and second line of ALK TKI treatment, with or without chemotherapy.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib + Alectinib | Crizotinib + Brigatinib | Crizotinib + Ceritinib | Alectinib + Brigatinib | Alectinib + Ceritinib | Alectinib + Lorlatinib | Ceritinib + Alectinib | Ceritinib + Brigatinib | Ceritinib + Lorlatinib | Crizotinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Chemotherapy | Alectinib + Brigatinib + Chemotherapy | Alectinib + Ceritinib + Chemotherapy | Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Chemotherapy | Ceritinib + Brigatinib + Chemotherapy | Ceritinib + Lorlatinib + Chemotherapy
Number analyzed (Participants) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of participants | 0.00 |  | 0.00 |  |  |  |  |  |  |  |  | 0.00 |  |  |  |  |  |

26. Primary Outcome: Percentage of Participants Alive After 6 Years From Index Date: Based on ALK Sequencing, 3 Lines of ALK TKI Treatment
Description: Participants alive after six years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure OS was reported for participants who received 3 lines of ALK inhibitor treatment. Reporting arms were based on type of first line ALK TKI treatment, second line of ALK TKI treatment, and third line of ALK TKI treatment, with or without chemotherapy.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib + Alectinib + Ceritinib | Crizotinib + Alectinib + Lorlatinib | Crizotinib + Alectinib + Brigatinib | Crizotinib + Ceritinib + Alectinib | Crizotinib + Ceritinib + Lorlatinib | Crizotinib + Ceritinib + Brigatinib | Crizotinib + Brigatinib + Alectinib | Crizotinib + Brigatinib + Lorlatinib | Alectinib + Brigatinib + Lorlatinib | Alectinib + Lorlatinib + Brigatinib | Alectinib + Lorlatinib + Ceritinib | Ceritinib + Alectinib + Lorlatinib | Ceritinib + Alectinib + Brigatinib | Crizotinib + Alectinib + Ceritinib + Chemotherapy | Crizotinib + Alectinib + Lorlatinib + Chemotherapy | Crizotinib + Alectinib + Brigatinib + Chemotherapy | Crizotinib + Ceritinib + Alectinib + Chemotherapy | Crizotinib + Ceritinib + Lorlatinib + Chemotherapy | Crizotinib + Ceritinib + Brigatinib + Chemotherapy | Crizotinib + Brigatinib + Alectinib + Chemotherapy | Crizotinib + Brigatinib + Lorlatinib + Chemotherapy | Alectinib + Brigatinib + Lorlatinib + Chemotherapy | Alectinib + Lorlatinib + Brigatinib + Chemotherapy | Alectinib + Lorlatinib + Ceritinib + Chemotherapy | Ceritinib + Alectinib + Lorlatinib + Chemotherapy | Ceritinib + Alectinib + Brigatinib + Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of participants |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.00 |  |  |  |  |  |  |  |  |

27. Primary Outcome: Percentage of Participants Alive After 6 Years From Index Date: Based on ALK Sequencing, More Than or Equal to (>=) 4 Lines of ALK TKI Treatment
Description: Participants alive after six years from index date (date of first ALK TKI prescription) to the date of death due to any cause or censoring date (latest available date in data), were reported. In this outcome measure, data is reported for participants who received >=4 lines of ALK inhibitor treatment with or without chemotherapy.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Number; unit: Percentage of participants
Arm/Group | >=4 Lines of ALK TKI | >=4 Lines of ALK TKI With Chemotherapy
Number analyzed (Participants) | 1 | 3
Percentage of participants | 0.00 | 33.33

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events not collected during the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met; hence, adverse events were not collected and reported.
Arm/Group | Participants With No First Line Chemotherapy | Participants With First Line Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to ethical compliance study team ensured results would not be reported for those cohorts/groups which had less than 5 participants at the index date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT04647110/Prot_SAP_000.pdf